CLINICAL TRIAL: NCT01568177
Title: Cardiac Autonomic Function in Women with Microvascular Coronary Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22264
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Microvascular Coronary Dysfunction
Keywords: MCD
MeSH Terms: conditions — Macular dystrophy, corneal type 1 | interventions — technetium tc-99m tetrofosmin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (3):
- abnormal CRT (Other): 40 subjects with microvascular coronary dysfunction (MCD) defined as abnormal CRT.
  Visits 1, 2, and 3
  Interventions: Behavioral: Mental Stress Testing; Other: Peripheral Arterial Tonometry (PAT) Testing; Other: Heart Rate Variability (HRV); Other: RESPeRATE Breathing Trial; Procedure: SPECT cardiac scan with 123I-mIBG and Myoview
- Cardiac Syndrome X (Other): 20 subjects with symptoms and normal stress tests, no MCD. Visits 1 and 2
  Interventions: Behavioral: Mental Stress Testing; Other: Peripheral Arterial Tonometry (PAT) Testing; Other: Heart Rate Variability (HRV); Other: RESPeRATE Breathing Trial; Procedure: SPECT cardiac scan with 123I-mIBG and Myoview
- normal reference controls (Other): 40 normal reference controls subjects Visits 1 and 2
  Interventions: Behavioral: Mental Stress Testing; Other: Peripheral Arterial Tonometry (PAT) Testing; Other: Heart Rate Variability (HRV); Other: RESPeRATE Breathing Trial; Procedure: SPECT cardiac scan with 123I-mIBG and Myoview

INTERVENTIONS:
Behavioral: Mental Stress Testing — Mental stress testing is used to test the mechanistic pathways through which biobehavioral variables are involved in the pathogenesis of MCD in women.
Other: Peripheral Arterial Tonometry (PAT) Testing — PAT measurements will be used to predict ischemia in patients with MCD. PAT will be measured by Endo PAT 2000 (Itamar® Medical Ltd).
Other: Heart Rate Variability (HRV) — Holter monitor will be used to measure heart rate and rhythm for approximately 24 hours.
Other: RESPeRATE Breathing Trial — RESPeRATE Breathing will test whether a controlled breathing relaxation technique using an FDA-approved paced breathing device, RESPeRATE, helps with chest pain and shortness of breath and will test to see if this form of biofeedback or relaxation technique helps with heart rate variability during mental stress.
Procedure: SPECT cardiac scan with 123I-mIBG and Myoview — Single Photon Emission Computed Tomography (SPECT) cardiac scan with 123I-mIBG and Myoview will be used to measure cardiac sympathetic activity.

SUMMARY:
Microvascular coronary dysfunction (MCD) (abnormities in small blood vessels/arteries in heart) with symptoms of persistent chest pain impacts women. There are an estimated 2-3 million women in the US with MCD and about 100,000 new cases annually. Autonomic nervous system (ANS) is part of the central nervous system to help people adapt to changes in their environment. It controls what are normally involuntary activities, such as heart rate, respiration (breathing), body temperature, blood pressure, and urinary function. However, there is a limited understanding of the role of ANS in MCD. This research is proposed to investigate cardiovascular reactivity to mental stress and the cardiac (heart) nervous system in women with MCD using mental stress testing, peripheral vascular testing, advanced cardiac imaging and cardiac autonomic function testing. 100 participants will be recruited in the next five years.

DETAILED DESCRIPTION:
There are three groups in this study: 40 MCD subjects with abnormal coronary reactivity testing (CRT), 20 CSX subjects with symptoms and nomral stress testing, and 40 normal controls. Normal controls will complete two study visits while MCD subjects may have up to three study visits.

Recruiting participants from Protocol 14906:

To date, no participants from Protocol 14906 have completed the study yet. All the participants who are currently enrolled in 14906 will be approached by the investigator at their next study visits. Prospectively new participants will be approached while they are consented for 14906.

Recruiting participants from Protocol 11753:

Participants who are currently enrolled in Protocol 11753 will be approached at their next study visits. Prospectively new participants will be approached while they are consented for 11753. Research staff may also identify past patients who have completed 11753 and fulfill the requirements for healthy individuals.

All participants will be asked to undergo research procedures including mental stress tasks, heart rate variability, cold pressor testing, and peripheral arterial tonometry. These procedures are described below by visit:

VISIT ONE:

MENTAL STRESS TESTING Mental Stress Testing will be used to study what happens to heart rate, blood pressure, heart rhythm, and blood vessels in arms and hands when participants are in a stressful situation. It will take up to 3 hours to complete all the procedures in the mental stress testing including the following specific procedures: In Mental Stress Tasks, different types of stress testing, including a speech task over a situation that made participants upset or angry, and/or a math test involving adding or subtracting numbers under a specific constraint, and/or a memory test, will be administered to study the effect of stress on heart; In Heart Rate Variability (HRV), participants will be asked to wear a Holter monitor that measures heart rate and rhythm for approximately 24 hours; In Cold Pressor Testing, participants' heart rate, blood pressure, heart rhythm, and blood vessels will be monitored; In Peripheral Arterial Tonometry (PAT), a blood pressure cuff will be placed on one arm and probes will be placed on participants' fingers. The probes and cuff are attached to a monitoring device that transfers a waveform graph of participants' pulse. Then the blood pressure cuff will be inflated for 5 minutes. At the end of the 5-minute period, the blood pressure cuff will be deflated to get the final tracings.

RESPERATE BREATHING TRIAL In subjects who have MCD, to know whether a controlled breathing relaxation technique using an FDA-approved paced breathing device, RESPeRATE, helps with chest pain and shortness of breath and to test to see if this form of biofeedback or relaxation technique helps with heart rate variability during mental stress, MCD subjects will be randomized to completing a RESPeRATE breathing trial or performing their own choice of relaxation technique for 8 weeks.

VISIT TWO:

SINGLE PHOTON EMISSION COMPUTED TOMOGRAPHY (SPECT) CARDIAC SCAN WITH 123I-MIBG AND MYOVIEW Single Photon Emission Computed Tomography (SPECT) cardiac scan with 123I-mIBG and Myoview will be used to measure cardiac sympathetic activity. The test will take approximately 5 hours with approximately 3.5 hours of break in the middle.

VISIT THREE:

REPEATED MENTAL STRESS TESTING Only subjects with MCD will have the visit that will take about 3 hours to complete. During this visit, MCD subjects will be asked to complete repeated Mental Stress Testing, including Mental Stress Tasks, Holter Heart Rate Variability, and PAT testing as outlined above

All the procedures are research-related. Participants may consent to some but not all of the procedures due to our current limited funding.

There are no collaborations with other sites.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Protocol 14906:

* Women with symptomatic angina or angina equivalent;
* Age > 18 yrs old;
* No obstructive CAD at coronary angiography (performed within the previous 24 months);
* Competent to give informed consent.

Inclusion criteria for Protocol 11753:

* Women without signs and symptoms of myocardial ischemia (chest pain, abnormal stress testing, abnormal noninvasive testing);
* No cardiac risk factors by Framingham/NCEP criteria;
* Age (35-65) matched to the WISE MCD population;
* A normal maximal exercise stress test.

Exclusion Criteria:

Exclusion criteria for Protocol 14906:

* Obstructive CAD greater than or equal to 50% luminal diameter stenosis in greater than or equal to 1 epicardial coronary artery;
* Acute coronary syndrome (defined by the ACC/AHA criteria, Braunwald 2000);
* Primary valvular heart disease clearly indicating the need for valve repair or replacement;
* Patients with concurrent cardiogenic shock or requiring inotropic or intra-aortic balloon support;
* Prior or planned percutaneous coronary intervention or CABG;
* Acute MI;
* Prior non-cardiac illness with an estimated life expectancy < 4 years;
* Unable to give informed consent;
* Chest pain with a non-ischemic etiology (e.g.,pericarditis, pneumonia, esophageal spasm);
* Contraindications to CMRI (e.g., AICD, pacemaker, untreatable claustrophobia or known angio-edema);
* Women with intermediate coronary stenoses (> 20% but < 50% luminal diameter stenosis assessed visually at the time of angiography) will undergo clinically indicated IVUS testing based on the judgement of the operator; Those determined to have flow-obstructing stenosis will be excluded from the overall study;
* Participation in a research study that conflicts with the current WISE study.
* Women with coronary stenosis ≥50% in any epicardial coronary artery, assessed visually at the time of angiography, will not be included in the CRT subgroup.
* Women who are pregnant.
* Males

Exclusion criteria for Protocol 11753:

* Contraindications to CMR testing (metal devices in chest, claustrophobia, known angioedema);
* Contraindication to Adenosine including asthma, heart block (second and third degree) and sinus node disease, significant COPD/asthma, or systemic hypotension (<90mmHg);
* Contraindication to Dobutamine including severe systemic hypertension (≥ 220/120 mmHg), unstable angina, significant aortic valve stenosis, complex cardiac arrhythmia including uncontrolled atrial fibrillation, hypertrophic obstructive cardiomyopathy, myocarditis, endocarditis, pericarditis, or uncontrolled congestive heart failure;
* Contraindication to Gadolinium (renal impairment);
* Any renal disease;
* Pregnant and lactating women;
* Inability to perform exercise, e.g. orthopedic limitations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-02; Primary Completion 2024-02 (Actual); Study Completion 2024-02 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Reactivity (CVR) | 24 hours
  Cardiovascular Reactivity (CVR)

CONTACTS AND LOCATIONS:
Overall Officials: C. Noel Bairey Merz, M.D., Principal Investigator — Cedars-Sinai Medical Center; Puja Mehta, M.D., Principal Investigator — Emory University
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes